CLINICAL TRIAL: NCT04757129
Title: Dynamic Changes of Circulatory and Respiratory Function After Thrombolysis in Patients With Acute Pulmonary Embolism
Brief Title: Changes of Cardiopulmonary Function After Thrombolysis in Patients With Pulmonary Embolism
Acronym: CCFATAPE
Status: Recruiting | Type: Observational
Sponsor: Bin He (Other)
Responsible Party: Sponsor-Investigator, Bin He, Attending physician of Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Other Study IDs: JSSRMYY-HB-2
Record Dates: First submitted 2021-01-29; First posted 2021-02-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Acute Pulmonary Embolism
Keywords: acute pulmonary embolism; thrombolysis; Alteplase; cardiopulmonary function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thrombolysis success group: Echocardiography was performed 48 hours after thrombolysis to evaluate the success of thrombolysis according to previous report.
- thrombolysis failure group: Echocardiography was performed 48 hours after thrombolysis to evaluate the success of thrombolysis according to previous report.

SUMMARY:
The investigators expect to enroll about 80-100 acute pulmonary embolism patients treated with thrombolysis in two hospitals. Dynamic changes of cardiopulmonary function after thrombolysis are detected to evaluate which indicators can quickly reflect the effectiveness of thrombolysis.

DETAILED DESCRIPTION:
About 80-100 acute pulmonary embolism(APE) patients treated with thrombolysis are enrolled in the First Affiliated Hospital with Nanjing Medical University and Nanjing Drum Town Hospital from January 1, 2020, to June 30, 2024. According to the 2019 ESC guideline, the standards for thrombolysis in APE patients are as follows: within 2 weeks of onset; high-risk pulmonary embolism; medium-high-risk pulmonary embolism with symptoms of aggravation.

Investigators dynamically monitor cardiopulmonary function of participants after thrombolysis, including blood pressure, heart rate, respiratory rate, blood gas analysis, 2-dimensional echocardiography (left and right ventricular diameter, pulmonary artery pressure, interventricular septum) and laboratory tests (cTnT,pro-BNP).participants are divided into two groups: thrombolytic success group and thrombolytic failure group according the previously reported criterion which is evaluated 48h after thrombolysis.

Cardiopulmonary characteristics are analyzed to seek accurate and rapid index to reflect success of thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* medium-high risk or high risk pulmonary embolism and treated with thrombolysis

Exclusion Criteria:

* lack of radiologic evidence to diagnose APE
* death within 48 hours after thrombolytic therapy
* unable to partner treatment and leaving hospitals
* missing other necessary data
* pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: medium-high risk or high risk pulmonary embolism and treated with thrombolysis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
cardiopulmonary function changes | 48 hours after thrombolysis
  changes of PO2，SBP，HR, cardiac ultrasound index and vasoactive drug dosage

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China